CLINICAL TRIAL: NCT03094793
Title: Impact of Interictal Electroencephalographic Abnormalities on the Stability of Attention in the Epilepsies in Adults and Children
Brief Title: Impact of Interictal Electroencephalographic Abnormalities on the Stability of Attention in the Epilepsies
Acronym: COGNIT-AIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC14.374
Record Dates: First submitted 2016-08-16; First posted 2017-03-29 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy
Keywords: abnormal EEGs (AIC)
MeSH Terms: conditions — Epilepsy; Aicardi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- abnormal EEGs (Experimental)
  Interventions: Other: abnormal EEGs

INTERVENTIONS:
Other: abnormal EEGs — This study consists in a scalp EEG to detect, in real time, based on measurements of reaction time and accuracy of responses (recorded every two seconds), the level of attention given by the participant in a repetitive task of constant difficulty and correlate the behavioral results to AIC identified on the EEG recording. A computer equipped for the realization of the STABILO test is already available, its connection / synchronization with standard acquisition systems EEG data is already effective through an RS232 serial port.
  Included patients will see their EEG extended for fifteen minutes, during which they will carry out a computerized attentional task to evaluate the stability of the attention.
  Other Names: AIC

SUMMARY:
Cognitive disorders are a major problem in patients with epilepsy. One hypothesis is that the anomalies EEGs (AIC) may be responsible for short periods of attentional fluctuations causing a reduction of intellectual efficiency of patients. In this project, we propose to evaluate the impact of AIC on cognitive performance, specifically on attentional performance (central parameter of cognitive functioning) through the use of a computerized cognitive test (called STABILO, detailed below after) to measure, with good temporal sampling, the level of attentional engagement of patients in relation to their EEG activity.

The originality of this study lies in the synchronization of two examinations usually made independently (EEG and psychometric testing), respecting a precise temporal coupling. The aim is to provide clinicians with a tool to assess very quickly attentional fluctuations in epileptic patients, and to assess the potential impact of AIC on the occurrence of these changes, with possible therapeutic implications (treatment of AIC and / or specific treatment of attention deficit disorder).

The main objective of this study is to assess whether the presence of AIC EEG can induce a weakening of attentional performance.

DETAILED DESCRIPTION:
Cognitive disorders are a major problem in patients with epilepsy. A hypothesis supported by several authors postulated that abnormal EEGs (AIC) may be responsible for short periods of attentional fluctuations causing a reduction of intellectual efficiency of patients. Indeed, attention is a central parameter of human cognition, conditioning performance and welfare in virtually all areas of activity.

In this project, we propose to evaluate the impact of AIC on cognitive performance, specifically on attentional performance (central parameter of cognitive functioning) through the use of a computerized cognitive test (called STABILO, detailed below after) to measure, with good temporal sampling, the level of attentional engagement of patients in relation to their EEG activity.

The originality of this study lies in the synchronization of two examinations usually made independently (EEG and psychometric testing), respecting a precise temporal coupling. The aim is to provide clinicians with a tool to assess very quickly attentional fluctuations in epileptic patients, and to assess the potential impact of AIC on the occurrence of these changes, with possible therapeutic implications (treatment of AIC and / or specific treatment of attention deficit disorder).

This study consists in a scalp EEG to detect, in real time, based on measurements of reaction time and accuracy of responses (recorded every two seconds), the level of attention given by the participant in a repetitive task of constant difficulty and correlate the behavioral results to AIC identified on the EEG recording. A computer equipped for the realization of the STABILO test is already available, its connection / synchronization with standard acquisition systems EEG data is already effective through an RS232 serial port.

Included patients will see their EEG extended for fifteen minutes, during which they will carry out a computerized attention task (This is the STABILO experimental protocol developed by JP Lachaux and V. Herbillon) allowing the evaluation of the stability of 'attention.

ELIGIBILITY:
Inclusion Criteria:

* Patient major or minor age 6 to 65 (L1121-7 CSP)
* Written agreement of participation in the study patient and his legal representative
* Epilepsy proved, during diagnosis, or TDA justifying the realization of an EEG or video-EEG monitoring

Exclusion Criteria:

* Patient deprived of liberty by a judicial or administrative decision (L1121-6 CSP)
* Major Patients undergoing a legal protection measure or unable to consent (L1121-8 CSP)
* Pregnant or lactating women (L1121-5 CSP)
* Handicap making it impossible to complete the test (severe intellectual disability, severe motor deficit of the upper limbs, blindness)

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Presence of AIC measured by an EEG on attentional performance | 15 minutes
  Effect of AIC on attentional fluctuations

CONTACTS AND LOCATIONS:
Overall Officials: Philippe KAHANE, MD, PUPH, Principal Investigator — pkahane@chu-grenoble.fr
Locations (2):
- France (2):
  - University Hospital Grenoble, Grenoble
  - HCL, Lyon

IPD SHARING:
Plan to Share IPD: No